CLINICAL TRIAL: NCT06827353
Title: Retrospective Study to Evaluate Niraparib Versus Bevacizumab as Maintenance Therapy After First-line Treatment With Platinum-based Chemotherapy in Patients With de Novo Ovarian Cancer Without Homologous Recombination Deficiency
Brief Title: Niraparib Versus Bevacizumab as Maintenance Therapy in Patients With de Novo Ovarian Cancer Without Homologous Recombination Deficiency
Acronym: OVNI-B
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 24.10.24
Record Dates: First submitted 2024-11-05; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian cancer; Epithelial carcinoma; BRCA wild type; HRP; bevacizumab; niraparib; maintenance therapy; survival
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma | interventions — Maintenance; Bevacizumab; niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- niraparib: Patients who received niraparib as maintenance therapy
  Interventions: Drug: maintenance therapy with niraparib
- bevacizumab: Patients who received bevacizumab as maintenance therapy
  Interventions: Drug: maintenance therapy with bevacizumab

INTERVENTIONS:
Drug: maintenance therapy with bevacizumab — Maintenance therapy after platine-based chemotherapy in non-mutated advanced ovarian cancer is unclear. Arm of patients that received bevacizumab after chemotherapy.
  Other Names: bevacizumab; niraparib
  Groups: bevacizumab
Drug: maintenance therapy with niraparib — Maintenance therapy after platine-based chemotherapy in non-mutated advanced ovarian cancer is unclear. Arm of patients that received niraparib after chemotherapy.
  Groups: niraparib

SUMMARY:
Background: High-grade serous epithelial ovarian cancer is a disease with a poor prognosis in the advanced stages (stages III and IV). For patients with no biomolecular abnormalities, there are two maintenance treatments available after first-line chemotherapy: bevacizumab or niraparib. There is no prospective or strong retrospective study comparing these two therapies.

Hypothesis: Patients receiving bevacizumab are different from those receiving niraparib.

Objective: To compare the progression-free survival (PFS) of patients with high-grade stage III and IV ovarian carcinoma who received chemotherapy with those who received maintenance treatment with bevacizumab and those who received niraparib.

Method: Retrospective, multicenter study based on data collected from the patient's medical record. Eligible patients are all patients diagnosed with de novo high-grade serous epithelial ovarian carcinoma who have received first-line platinum-based chemotherapy followed by maintenance treatment with bevacizumab or niraparib. All eligible patients will be included. Patients with a BRCA mutation and/or a positive HRD score will be excluded. Data will be collected using an electronic CRF. The inclusion period is from October 2020 to December 2023.

DETAILED DESCRIPTION:
Introduction The incidence of ovarian cancer in France is estimated at over 5,100 cases/year in 2018. The most common histological form is high-grade serous epithelial carcinoma, which accounts for around 70% of ovarian cancers. Mortality is estimated at over 3,400 cases per year. The management of newly-diagnosed patients is based on multimodal treatment with maximal cytoreductive surgery, platinum-based chemotherapy and targeted therapy. For patients with advanced disease (stage III or IV), peri-operative or adjuvant chemotherapy with carboplatin combined with paclitaxel is the standard of treatment. At the end of this treatment, patients benefit from maintenance therapy, which may differ according to their biomolecular characteristics. For patients with a BRCA gene mutation or a high HRD score, the standard treatment is a combination of poly-ADP-ribose-polymerase inhibitor (iPARP) and an anti-VEGF antiangiogenic, bevacizumab.

On the other hand, for patients with no BRCA mutation or with a low HRD score (known as HRP), there are two treatment standards. They can be treated with an iPARP, niraparib. Indeed, the phase III PRIMA trial, which evaluated survival in patients with advanced ovarian cancer regardless of BRCA or HRD status, showed an improvement in progression-free survival (PFS) on an intention-to-treat basis. However, in the population of patients without BRCA and HRP mutations, PFS was 8.1 months in the niraparib group versus 5.4 months in the placebo group. The difference was statistically significant, with a hazard ratio of 0.68 (95% confidence interval 0.49-0.94). Overall survival data were not yet mature in 2023 in the most recent publication.

These same patients may also benefit from maintenance treatment with bevacizumab. A benefit in terms of PFS and OS has been demonstrated for populations at high risk of relapse (stage IV, or non-operable stage III or non-maximal surgery) in the ICON7 phase III study. In the GOG-0218 phase III study, bevacizumab was only shown to benefit progression-free survival.

Thus, both therapeutic strategies can be proposed as maintenance treatment after first-line chemotherapy for patients with advanced high-grade epithelial ovarian carcinoma in the non-mutated BRCA and HRP subpopulation. The data available to help choose between the two molecules are limited. The safety profile of each molecule and the contraindications may help in the choice. In their absence, there are no validated criteria in the scientific literature. The KELIM score (CA-125 ELIMination of Rate Constant K) can be used to predict iPARP efficacy. However, it has not been validated in this indication, since it was originally developed to predict chemosensitivity in these patients. Finally, there are no studies directly comparing the efficacy of bevacizumab with niraparib in this population.

Real-life data are therefore needed to understand and analyze prescribing practices, in order to identify avenues to aid therapeutic choice. Our study therefore aims to describe a population of patients with advanced high-grade epithelial ovarian carcinoma treated with maintenance bevacizumab or niraparib after platinum-based chemotherapy.

Study aim

Main objective:

To compare the progression-free survival (PFS) of patients with high-grade stage III and IV epithelial ovarian carcinoma who received chemotherapy between those who received maintenance treatment with bevacizumab and those who received niraparib.

Secondary objectives A. To describe the OS of the two groups. B. To compare the clinical, biological and sociodemographic characteristics of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* De novo diagnosis of stage III or IV high-grade epithelial ovarian carcinoma, not candidate for primary tumor reduction surgery.
* De novo diagnosis of high-grade epithelial ovarian carcinoma benefiting from a combination of chemotherapy and maximal cytoreduction surgery
* All patients who have received maintenance treatment after chemotherapy with bevacizumab or niraparib monotherapy.

Exclusion Criteria:

* Disease progression after chemotherapy
* Presence of a BRCA mutation (somatic or germline)
* Positive HRD score

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Identification of eligible patients in each center will be selected using the following criteria:
  * Ovarian cancer
  * Stage III or stage IV
  * Treatment initial surgery followed by chemotherapy or initial chemotherapy
  * Maintenance treatment with targeted therapy Then, inclusion and exclusion criterias will be applied . An electronic CRF (RedCap) will be used for data records.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival of patients with high-grade stage III and IV epithelial ovarian carcinoma who received chemotherapy between those who received maintenance treatment with bevacizumab and those who received niraparib. | From date of maintenance therapy start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 38 months
  Progression-free survival (PFS) defined as the time from initiation of maintenance therapy with bevacizumab monotherapy or niraparib to the date of disease progression or death from any cause. Disease progression is defined as cessation of maintenance therapy due to radiological and/or biological progression at the discretion of the oncologist managing the patient.

SECONDARY OUTCOMES:
Overall survival of the two groups | From date of maintenance therapy start until the date of death from any cause, assessed up to 38 months
  Overall survival (OS) defined as time from initiation of maintenance therapy with bevacizumab monotherapy or niraparib to date of death from any cause

OTHER OUTCOMES:
CA-125 ELIMination rate constant K (KELIM) score between groups | From date of randomization until the date of death from any cause, whichever came first, assessed up to 38months
  If CA-125 ELIMination rate constant K (KELIM) score result is less than value 1 patients will be classified as unfavorable risk. If KELIM score result equal or more than 1, patients will be classified as favorable risk.
Radiological response | From date of maintenance therapy start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 38 months
  Radiologic response according on CT-scan after chemotherapy, at maintenance therapy will be adressed using the Response Evaluation Criteria In Solid Tumours version 1.1 as fur categories : progression disease, stable disease, partial response disease and complete response disease
Comparrative performans status between two groups | From date of maintenance therapy start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 38 months
  Performance status Eastern Cooperative Oncology Group (PS ECOG) scalled from 0 to 5. Score 0 correspond to fully active, able to carry on all pre-disease performance without restriction. Score 5 correspond to Dead patient.
Quality of surgical resection | From date of maintenance therapy start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 38 months
  This issue will be addressed using the pathologist and the residual tumor (R) classification. R0 corresponds to resection for cure or complete remission. R1 to microscopic residual tumor, R2 to macroscopic residual tumor

CONTACTS AND LOCATIONS:
Overall Officials: soufyan annakib, M.D., Principal Investigator; Frédéric Fiteni, M.D., Ph.D., Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, Occitanie, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be available only on demande. Available data will be only those used for study results publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After results publication.
Access Criteria: Only on demande.

REFERENCES:
- [Background] Hannaway N, Kassaris S, Davies JM, Smrke A, Tinker A, Drew Y. Using chemotherapy response by KELIM score to predict response to first line maintenance PARP inhibitor therapy in non-BRCA mutant/homologous recombination deficiency (HRD) unknown high grade serous ovarian cancer (HGSOC). J Clin Oncol. 1 juin 2023;41(16_suppl):e17547-e17547.
- [Background] Burger RA, Brady MF, Bookman MA, Fleming GF, Monk BJ, Huang H, Mannel RS, Homesley HD, Fowler J, Greer BE, Boente M, Birrer MJ, Liang SX; Gynecologic Oncology Group. Incorporation of bevacizumab in the primary treatment of ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2473-83. doi: 10.1056/NEJMoa1104390. PMID 22204724
- [Background] Gonzalez-Martin A, Pothuri B, Vergote I, DePont Christensen R, Graybill W, Mirza MR, McCormick C, Lorusso D, Hoskins P, Freyer G, Baumann K, Jardon K, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Lund B, Backes F, Barretina-Ginesta P, Haggerty AF, Rubio-Perez MJ, Shahin MS, Mangili G, Bradley WH, Bruchim I, Sun K, Malinowska IA, Li Y, Gupta D, Monk BJ; PRIMA/ENGOT-OV26/GOG-3012 Investigators. Niraparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2391-2402. doi: 10.1056/NEJMoa1910962. Epub 2019 Sep 28. PMID 31562799
- [Background] Gonzalez-Martin A, Harter P, Leary A, Lorusso D, Miller RE, Pothuri B, Ray-Coquard I, Tan DSP, Bellet E, Oaknin A, Ledermann JA; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Newly diagnosed and relapsed epithelial ovarian cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Oct;34(10):833-848. doi: 10.1016/j.annonc.2023.07.011. Epub 2023 Aug 17. No abstract available. PMID 37597580
- [Background] Defossez G, le Guyader-Peyrou S, Uhry Z. Estimations nationales de l'incidence et de la mortalité par cancer en France métropolitaine entre 1990 et 2018. Saint-Maurice (Fra): Santé publique France; 2019.